CLINICAL TRIAL: NCT06604364
Title: realtà Aumentata Generatrice di Ansia Zero
Brief Title: Virtual Reality for Reducing Anxiety in Pediatric Orthopedic Surgery
Acronym: RAGAZ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 211/2024/DISP/IOR
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Virtual Reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control (No Intervention): pre-surgery sedation
- VR (Experimental): virtual reality sedation
  Interventions: Device: hypno VR

INTERVENTIONS:
Device: hypno VR — pre-surgery sedation using virtual reality headset
  Arms: VR

SUMMARY:
This study, titled "R.A.G.A.Z.: Virtual Reality for Reducing Anxiety and Pain in Pediatric Orthopedic Surgery," aims to see if using virtual reality (VR) can help children feel less anxious and experience less pain during minor orthopedic surgeries. The research will compare the effects of VR to the usual pre-surgery sedative medication.

**Study Hypotheses**

The researchers hypothesize that using VR will:

1. Reduce anxiety levels in children before and after surgery compared to standard sedative medication.

**Who can participate?**

* Children aged 7 to 12 years
* Undergoing minor orthopedic surgery lasting less than 60 minutes
* Eligible for regional anesthesia

**Study Process**

Participants will be randomly assigned to one of two groups:

1. VR Group: Children will use VR headsets to immerse themselves in calming virtual environments before and during the surgery.
2. Standard Care Group: Children will receive standard sedative medication before surgery.

The study will measure:

* Levels of anxiety before and after surgery using a specific anxiety meter (CAM-S).
* Stress hormone levels (cortisol, adrenaline, noradrenaline) from blood samples.
* Pain levels at different times after surgery.
* How well children cooperate during medical procedures.
* Satisfaction levels of children, parents, and surgeons.

The study is being conducted by IRCCS - Istituto Ortopedico Rizzoli in Bologna, Italy. It is a non-profit study funded by donations.

The goal is to find out if VR can reduce the need for sedatives, decrease anxiety and pain, and improve the overall surgical experience for children.

DETAILED DESCRIPTION:
**Detailed Description**

This study, titled "R.A.G.A.Z.: Virtual Reality for Reducing Anxiety and Pain in Pediatric Orthopedic Surgery," aims to evaluate the effectiveness of virtual reality (VR) in reducing perioperative anxiety and pain in children undergoing minor orthopedic surgeries. The study will compare the use of VR headsets to the traditional method of pre-surgery sedation with medication.

**Purpose of the Study**

The primary objective of this study is to determine whether VR can provide better control of anxiety in pediatric patients before and after anesthetic and surgical procedures. The study will also assess whether VR can reduce the need for sedative and pain-relief medications, thereby minimizing potential side effects and improving recovery times.

**Study Hypotheses**

The researchers hypothesize that VR will:

1. Significantly reduce anxiety levels in children before and after surgery compared to standard sedation practices.
2. Lower stress hormone levels (cortisol, adrenaline, noradrenaline) associated with surgical procedures.
3. Reduce the perceived pain during and after surgery.
4. Decrease the overall consumption of sedative and analgesic medications.
5. Good patient compliance during medical procedures.
6. Good satisfaction levels for patients, their parents, and healthcare providers.

**Study Design**

This is a non-profit, randomized controlled trial conducted at the IRCCS - Istituto Ortopedico Rizzoli in Bologna, Italy. The study will include 50 children aged 7 to 12 years, who are candidates for minor orthopedic surgeries lasting less than 60 minutes. Participants will be randomly assigned to one of two groups:

1. **VR Group**: Children in this group will use VR headsets to experience calming virtual environments such as underwater scenes or peaceful gardens. The VR sessions will begin before the surgical procedure and continue through the perioperative period.
2. **Standard Care Group**: Children in this group will receive the usual care, which includes pre-surgery sedation with midazolam, a common sedative used to reduce anxiety.

**Procedures**

* **Anxiety Assessment**: The Children's Anxiety Meter-State (CAM-S) will be used to measure anxiety levels at multiple points: preoperatively, upon arrival at the operating room, and at 3, 6, and 24 hours postoperatively.
* **Stress Hormone Levels**: Blood samples will be taken at the time of venipuncture to measure cortisol, adrenaline, and noradrenaline levels, which are indicators of surgical stress.
* **Pain Assessment**: Pain levels will be evaluated using the Faces Pain Scale-Revised (FPS-R) at various postoperative intervals (3, 6, and 24 hours).
* **Patient Compliance**: The Modified Induction Compliance Checklist (MICC) will be used to assess how well children comply with medical procedures such as venipuncture and anesthesia administration.
* **Satisfaction Surveys**: Satisfaction levels of patients, parents, and surgeons will be recorded using a scale from 1 to 10. This will assess overall satisfaction with the VR intervention and the surgical experience.

**Expected Outcomes**

The study aims to demonstrate that VR can effectively reduce perioperative anxiety and pain, leading to a lower requirement for sedatives and analgesics. By providing a non-pharmacological method to manage anxiety and pain, VR could improve the overall surgical experience for pediatric patients and enhance recovery outcomes. Additionally, the study seeks to validate the feasibility and acceptability of VR as a standard practice in pediatric surgical settings.

**Study Timeline**

The study is expected to last 24 months, including patient enrollment, data collection, and analysis. Each participant will be involved from the preoperative visit through the first 24 hours post-surgery. The results will be analyzed and published to contribute to the growing body of evidence supporting the use of VR in medical procedures.

**Ethical Considerations**

The study will be conducted following the principles of the Declaration of Helsinki and Good Clinical Practice (GCP) guidelines. Informed consent will be obtained from all participants and their parents or guardians. The privacy and confidentiality of all participants will be strictly maintained.

This study has the potential to revolutionize the approach to managing perioperative anxiety and pain in pediatric patients, offering a safe, effective, and enjoyable alternative to traditional sedative medications.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7 to 12 years.
* Scheduled for minor orthopedic surgery with a duration of less than 60 minutes.
* Eligible for regional anesthesia.
* Able to understand and cooperate with the study procedures.
* Consent from both the child and their parent or legal guardian.

Exclusion Criteria:

* Facial trauma that prevents the use of VR headsets.
* Blindness or significant visual impairment.
* Deafness or significant hearing impairment.
* Cognitive impairments or intellectual disabilities.
* Inability to understand the language used in the VR content.
* Poor fit of the VR headset on the child's face.
* Inability to understand Italian.
* Current use of analgesics or sedatives at home.
* Certified psychiatric diagnosis.
* Epilepsy or history of seizures.
* Recent head trauma, severe headaches, or vertigo.
* Any condition deemed by the anesthesiologist to be unsafe for VR use.
* Failure to properly apply topical anesthetics before invasive procedures.
* Allergy to local anesthetics.
* Surgery duration expected to exceed 60 minutes.
* Anticipated need for general anesthesia or deep sedation requiring advanced airway management.
* Predicted difficult venous access (DIVA)

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06-03 (Estimated)

PRIMARY OUTCOMES:
anxiety level | 24 hours
  level of anxiety with cam-s

SECONDARY OUTCOMES:
hormons levels | preoperative
  levels of stress hormons
pain level | 24 hours
  difference in pain levels
compliance during induction | during induction
  compliance during induction of anesthesia with micc
drugs dosage | intraoperative
  dosage of drugs necessary for induction of anesthesia
surgeons satisfaction | immediately after the intervention
  general satisfaction of the surgeons from 1 to 10
parents satisfaction | immediately after the intervention
  general satisfaction of the parents from 1 to 10
or time occupation | intraoperative
  time of occupation of the or
adverse event | 24 hours
  adverse avent using virtual reality

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided